CLINICAL TRIAL: NCT07247201
Title: Phase 1/2 Trial Integrating Allogeneic NK Cells in High-risk Advanced Stage III-IV Nasopharyngeal Cancer Patients
Brief Title: Integrating Allogeneic NK Cells in High-risk Advanced Stage III-IV Nasopharyngeal Cancer Patients
Acronym: AlloNK1
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2024-2264; CSAINV22jul-0014 (Other Grant/Funding Number: National Medical Research Council (NMRC)); CTGIIT23jul-0003 (Other Grant/Funding Number: National Medical Research Council (NMRC))
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Carcinoma (NPC); Minimal Residual Disease; Recurrent Nasopharyngeal Carcinoma; Maximum Tolerated Dose
Keywords: Advanced Nasopharyngeal Cancer; Epstein-Barr Virus DNA; Allogeneic NK Cells; Maximum Tolerated Dose
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Concurrent and adjuvant allogeneic NK cell therapy (Experimental): Participants will receive standard chemoradiotherapy for locally advanced nasopharyngeal carcinoma along with adjuvant therapy of NK cells. Nk cells would be enriched and expanded using PBMCs from healthy donors.
  Phase 1 dose escalation study which uses 5 different dosages of 0.5 x 10^7, 0.8x10^7, 1.1x10^7, 1.4 x 10^7, and 1.8x10^7 to determine the Maximum tolerated dose (MTD). If the MTD is determined in phase 1, the study will enter phase 2, where the determined dose level will be used for participants. The participants will receive six intravenous NK cell infusions at weeks 3,6,7,8,9, and 10 during and after CRT. If the participant's EBV level is still detectable, they would be suggested for supplementary NK cell treatments for an additional four weeks.
  Interventions: Biological: Allogenic expanded Natural Killer Cells (AlloNK1)

INTERVENTIONS:
Biological: Allogenic expanded Natural Killer Cells (AlloNK1) — The NK cells would be enriched and expanded ex vivo in a GMP facility from healthy donor PBMCs. Prior to administration, the NK cells would be formulated in an infusion medium based on the corresponding dose level that is required for each participant.
  Participants will receive an intravenous infusion of NK cells during and after the standard CRT. Six doses are administered at weeks 3,6,7,8,9, and 10. In Phase 1, NK cell doses range from 0.5x10^7 to 1.8x10^7 cells/kg for the determination of the maximum tolerated dose (MTD). In phase 2, all participants will receive NK cells at the established MTD.

SUMMARY:
This clinical trial aims to determine whether Natural Killer (NK) cell therapy administered in combination with concurrent chemoradiotherapy (CRT) can reduce recurrence in patients with advanced nasopharyngeal cancer (NPC), and to identify the highest safe and tolerable dose of allogeneic NK cells. Allogeneic NK cells, derived from healthy donors, have demonstrated good tolerability in cancer patients.

The primary research questions are:

1. What is the maximum tolerated dose (MTD) of allogeneic NK cells when administered with CRT in NPC patients?
2. Can the addition of allogeneic NK cells to standard CRT reduce the proportion of NPC patients with detectable plasma EBV-DNA from 30% to 10%?

Phase 1: Participants will receive one of five escalating doses of allogeneic NK cells with CRT to determine the MTD.

Phase 2: Participants will receive the established MTD NK dose together with CRT.

Participants will undergo regular safety monitoring, side-effect assessment, measurement of plasma EBV-DNA levels, and surveillance for disease recurrence.

DETAILED DESCRIPTION:
The investigator plans to enrol 31 newly diagnosed NPC patients with Stage III-IVA/B (T1-4, N1-3, M0) disease who are scheduled to receive standard-of-care treatment over an estimated 24-36-month period.

The clinical trial consists of a Phase 1 dose-escalation study followed by a single-arm Phase 2 study. In Phase 1, at least six participants will be treated at the MTD of allogeneic NK cells, after which an additional 25 participants are expected to be enrolled in Phase 2.

Phase 1 will use the Bayesian Model Averaging Continual Reassessment Method (BMA-CRM) to determine the MTD, evaluating five NK-cell dose levels of 0.5×10⁷, 0.8×10⁷, 1.1×10⁷, 1.4×10⁷, and 1.8×10⁷ cells/kg, with the starting dose set at 0.8×10⁷ cells/kg. Dose-limiting toxicity (DLT) is defined as Grade 3 to 5 toxicities per CTCAE criteria, and the target toxicity limit (TTL) is set at a maximum allowable DLT probability of 30%. Toxicity probability will be reassessed whenever a DLT occurs to determine whether it exceeds the TTL. If the cohort completes evaluation at a given dose level and the toxicity probability is within the TTL, dose escalation will proceed; however, if the toxicity probability exceeds the TTL, the dose will be rejected, and de-escalation will occur. When toxicity probability is low, accelerated escalation may be implemented.

Phase 1 will conclude once six participants have been treated at the designated MTD without developing Grade 3 to 5 toxicities; at that point, the MTD will be accepted. All participants in Phase 1 will receive standard NPC treatment combined with the NK-cell dose evaluated at the time of their enrollment.

Phase 2 is a single-arm study based on historical findings that approximately 25% to 30% of locally advanced NPC patients continue to exhibit detectable circulating EBV-DNA following standard CRT. The study hypothesizes that the addition of allogeneic NK cells will reduce this proportion to 10%.

All participants in Phase 2 will receive standard CRT along with NK-cell infusions administered once weekly during weeks 3, 6, 7, 8, 9, and 10. Interleukin-2 (200 U/mL) will be co-administered with NK cells in Plasma-Lyte 148 supplemented with 2% human serum albumin (HSA). The primary endpoint of Phase 2 is the reduction in the proportion of patients with detectable post-treatment circulating EBV-DNA. At week 9, if the participants' circulating EBV-DNA levels have decreased but remain detectable, they will receive an optional additional four NK-cell infusions during weeks 12 to 15.

The secondary endpoint is the improvement in survival and recurrence rates within 24 to 36 months compared with historical cohorts receiving standard treatment alone. NK cells will be generated from healthy-donor PBMCs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with NPC Stage III-IVA/B (T1-4, N1-3, M0)
* Able to tolerate convectional CRT
* Detectable EBV level at diagnosis
* Adequate organ function ANC ≥ 1500/µL Platelet count ≥ 100,000/µL Creatinine clearance ≥60ml/minute Total bilirubin ≤ 1.5 x upper limit normal (ULN) AST ≤ 2 x upper limit normal ALT ≤ 2 x upper limit normal
* ECOG performance status of 0-1

Exclusion Criteria:

* History of Autoimmune Disease or any condition resulting in immunocompromised state (e.g., Drug induced)
* ECOG performance status above or equal to 2
* Poor Organ Function
* Lactating or pregnant
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Determine the MTD of allogenic NK cells | From enrollment to the end of treatment at week 10
  The primary objective of this trial is to determine the MTD of allogeneic NK cells when used with concurrent CRT in advanced NPC patients.
The percentage of patients with detectable plasma EBV-DNA decreased to 10% post treatment | From day of enrollment to the end of treatment at week 10
  Primary endpoint is set at the percentage of patients with detectable post-treatment circulating EBV-DNA has decreased from 30% to 10%.

SECONDARY OUTCOMES:
Determine the patient survival and recurrence rate post-treatment | 24 to 36 months after the last treatment done at week 10
  Secondary endpoint is in determining the change in patient survival and recurrence rate within 24-36 months post-treatment under this new treatment regimen when compare with historic cohorts under standard treatments

CONTACTS AND LOCATIONS:
Overall Officials: Lim Chwee Ming, Principal Investigator — Singapore General Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT07247201/Prot_SAP_000.pdf
  • Informed Consent Form: For NPC patients (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT07247201/ICF_001.pdf
  • Informed Consent Form: For Healthy Donors (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT07247201/ICF_002.pdf